CLINICAL TRIAL: NCT00510965
Title: Ranibizumab in Choroidal Neovascularization (CNV) Due to Pseudoxanthoma Elasticum (PXE, Groenblad-Strandberg-Syndrome)
Brief Title: Ranibizumab to Treat Choroidal Neovascularization (CNV) in Patients With Pseudoxanthoma Elasticum (PXE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Collaborators: Novartis (Industry)
Responsible Party: University of Bonn, University of Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002ADE03; EudraCT number 2006-006233-49
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2011-08

CONDITIONS: Choroidal Neovascularization
Keywords: choroidal neovascularization; angioid streaks; pseudoxanthoma elasticum; Groenblad-Strandberg-Syndrome; therapy; ranibizumab; lucentis; Choroidal neovascularization in patients with PXE
MeSH Terms: conditions — Choroidal Neovascularization; Angioid Streaks; Pseudoxanthoma Elasticum | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Intravitreal injection ranibizumab

INTERVENTIONS:
Drug: Intravitreal injection ranibizumab — Monthly intravitreal injection of 0.5mg ranibizumab in one eye over one year
  Other Names: Lucentis

SUMMARY:
The purpose of the study is to investigate the efficacy of a new drug called ranibizumab in the treatment of choroidal neovascularization in underlying angioid streaks due to Pseudoxanthoma elasticum. 10 patients will receive monthly injections of the drug in one eye over a period of one year.

DETAILED DESCRIPTION:
Pseudoxanthoma elasticum (PXE) is a rare hereditary systemic disease affecting mainly the skin, eyes and the cardiovascular system. Commonly, complicating choroidal neovascularization (CNV) of the central retina lead to a severely decreased visual acuity in the course of the disease. Onset of the symptoms varies with the extend of the PXE-associated findings.

In the past there has been no effective treatment for the disease's ocular complications. Recent studies in a limited number of patients with CNV treated with intravitreal injections of bevacizumab, an antagonist targeting vascular endothelial growth factor (VEGF), have shown a preservation of function and regression of CNV. An increase of visual acuity was reported in a subset of patients. Bevacizumab is a humanized antibody of which ranibizumab is a fragment.

This trial is initiated in order to investigate the effect of ranibizumab on functional outcome measures such as preservation of visual acuity as well as morphological outcome measures such as regression of CNV in angiography.

The safety and tolerability of ranibizumab will be investigated as well. As it has been tested on large numbers of patients suffering from age-related macular degeneration with only rare significant side effects or adverse events being reported, a good safety profile is assumed.

The study is conducted in a non-randomized, uncontrolled prospective setting at one center.

Patients will receive monthly injections over a period of one year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of choroidal neovascularization in patients with pseudoxanthoma elasticum
* Age between 18-65 years
* Patient must be able to follow protocol
* Written informed consent
* Genetic diagnosis of pseudoxanthoma elasticum
* Best corrected visual acuity between 20/200 - 20/32 in the treated eye

Exclusion Criteria:

* Patients who do not fulfill the inclusion criteria
* Patients with other retinal vascular diseases such as diabetic retinopathy or venous occlusive disease
* Ocular surgery 3 months before study enrollment
* History of uncontrolled glaucoma
* Active intraocular inflammation or inflammation of the ocular adnexa
* Subfoveal fibrosis in the study eye
* Inability to follow study protocol
* Major surgery one month before study enrollment
* History of severe cardiovascular disease or history of stroke 6 months before study enrollment
* Allergies against the substances or components of the study medication
* Low anticipated compliance
* Patients who participated in clinical trials simultaneously or within the last 60 days
* Pregnancy, lactation, women that may become pregnant and don't use safe contraception
* Chronic alcohol- or drug abuse within the last year
* Lacking legal competence or language ability
* Neurologic diseases such as multiple sclerosis
* Need of concomitant medication that is not allowed in combination with ranibizumab
* Previous intravitreal therapy with anti-angiogenic substances in the study eye within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | one year

SECONDARY OUTCOMES:
Reading ability | one year
Changes in retinal thickness assessed by optical coherence tomography | one year
Changes in parafoveal leakage assessed by fluorescein angiography | one year
Quality of life | one year

CONTACTS AND LOCATIONS:
Overall Officials: Frank G. Holz, MD, Principal Investigator — University of Bonn, Department of Ophthalmology; Hendrik PN Scholl, MD, MA, Principal Investigator — University of Bonn
Locations (1):
- University of Bonn, Bonn, Germany

REFERENCES:
- [Derived] Finger RP, Charbel Issa P, Hendig D, Scholl HP, Holz FG. Monthly ranibizumab for choroidal neovascularizations secondary to angioid streaks in pseudoxanthoma elasticum: a one-year prospective study. Am J Ophthalmol. 2011 Oct;152(4):695-703. doi: 10.1016/j.ajo.2011.03.022. Epub 2011 Jun 25. PMID 21704964
- See also: Related Info — http://www.augenklinik.uni-bonn.de